CLINICAL TRIAL: NCT00521378
Title: A Single-Blind, Placebo-Controlled, Dose-Ranging Trial of Oral HDV-Insulin in Patients With Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Diasome Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: DP 01-2007-01
Record Dates: First submitted 2007-08-23; First posted 2007-08-27 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: Diabetes; Type 1 and Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A study designed to determine the appropriate doses of Oral HDV Insulin at meal times.

ELIGIBILITY:
Inclusion Criteria:

Patients must satisfy all of the following inclusion criteria to be included in the study:

1. be male or female between the ages of18 and 65 years, inclusive;
2. have a current diagnosis of type 2 DM, which is currently managed with oral hypoglycemic agents for at least 3 months;
3. have a current physical examination that reveals no clinically significant abnormalities;
4. have no clinically significant abnormalities in vital signs;
5. have a body mass index (BMI) <38;
6. have a glycosylated hemoglobin (HbA1c) > 8 and <12;
7. have a C-peptide level >3 ng/mL;
8. have a typical fasting blood glucose levels of < 200 mg/dl (+/- 25 mg/dl);
9. be available for the entire study period, and be able and willing to adhere to protocol requirements;
10. if female of childbearing potential, must be using a reliable form of birth control; and,
11. provide written informed consent prior to admission into the study.

Exclusion Criteria:

1. have a history or presence of significant cardiac, gastrointestinal, endocrine, neurological, liver, or kidney disease, or conditions known to interfere with the absorption, distribution, metabolism, or excretion of insulin;
2. have a history of drug or alcohol dependency or psychological disease;
3. have any clinically significant illness during the 4 weeks prior to admission into the study;
4. require regular use of medication that interferes with the absorption and/or metabolism of insulin;
5. recent use (within 48 hours) of medications that interfere with blood glucose analyses, i.e., mannose, acetaminophen, dopamine, and ascorbic acid, which are all reported to alter glucose-oxidase type blood glucose analytical methods;
6. use of Avandia or Actos for treating diabetes;
7. participation in a clinical trial or use of an investigational drug within 30 days prior to admission to this study;
8. use of MAO inhibitors or enzyme-inducing or enzyme-inhibiting agents (eg, phenobarbital or carbamazepine) within 30 days prior to admission to this study;
9. are pregnant or lactating; 10. have an episode of severe hypoglycemia with seizure or coma within the past year;

11. have a history of ketoacidosis;

12. have any acute illness within 2 weeks prior to Screening; or,

13. have elevated liver enzymes (ALT, AST, alkaline phosphatase) >1.5 times the upper limit of normal.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Have a current diagnosis of type 2 DM, which is currently managed with oral hypoglycemic agents for at least 3 months
Enrollment: 6 (Actual)
Dates: Start 2007-09-17 (Actual); Primary Completion 2007-10-06 (Actual); Study Completion 2007-10-06 (Actual)

PRIMARY OUTCOMES:
Dose response of postprandial plasma glucose to escalated doses of oral HDV-insulin | 3 weeks
  To determine the dose response of postprandial plasma glucose to escalating doses (increased daily) of Oral HDV-Insulin given as single doses before breakfast, lunch and dinner, in addition to the Diabetes Mellitus (DM) subject's regular oral type 2 therapy
Daily glucodynamic profile of Oral HDV-Insulin | 3 weeks
  To compare the daily glucodynamic profile of Oral HDV-Insulin over the treatment days

CONTACTS AND LOCATIONS:
Locations (1):
- San Antonio, Texas, United States